CLINICAL TRIAL: NCT06257186
Title: Investigating the Effect of Art Therapy on Women With Fear of Childbirth During Pregnancy: A Mixed Method Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Ang Mei Qi, Nurse Clinician, KK Women's and Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/2493
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Fear of Childbirth; Pregnancy Related; Anxiety and Fear; Anxiety; Fear
MeSH Terms: conditions — Anxiety Disorders | interventions — Art Therapy

STUDY DESIGN:
Intervention Model Description: A mixed-methods sequential explanatory design will be used. Phase one will be quasi-experimental study design, comparing women with FOC who received art therapy (experimental group) and women who received routine antenatal care (control group). A qualitative descriptive design will be used in phase two to explore the experiences of the participants who had art therapy for FOC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art Therapy (Experimental): Women in the experimental group will be offered a series of three to five art therapy sessions, depending on the participants' needs/preferences. The art therapy sessions will be given anytime after consent has been obtained till approximately 36 weeks of gestation. The art therapy sessions are in addition to routine antenatal care.
  Interventions: Other: Art Therapy
- Routine Antenatal Care (No Intervention): Women in the control group will receive routine antenatal care.

INTERVENTIONS:
Other: Art Therapy — Participants assigned to the Intervention (Art Therapy) arm will be offered a series of three to five art therapy sessions, depending on the participants' needs/preferences. The art therapy sessions will be given anytime after consent has been obtained till approximately 36 weeks of gestation. The Art Therapy is given in addition to routine antenatal care.
  Arms: Art Therapy

SUMMARY:
Childbirth is a multifaceted experience and could involve both positive and negative feelings. Feelings of limited capability in the face of childbirth may result in a condition termed as Fear of Childbirth (FOC), which contributes to significantly higher risks of birth complications resulting in psychological trauma. This study aims to examine the effects of Art Therapy (AT) on FOC, perceived maternal parental self-efficacy, postpartum maternal infant bonding and postpartum depression.

A mixed-methods sequential explanatory design will be used. Phase one will adopt a quasi-experimental study design. Women who are aged 21 and above, English literate and having a singleton pregnancy will be approached to fill in the Fear of Birth Scale (FOBS). Participants with FOBS score of 60 and above will be considered as having FOC and will be invited to participate in the AT intervention. Participants who are agreeable to receive AT will be recruited in the experimental group. Participants who declined to participate in AT will receive routine antenatal care (control group). Outcomes that will be measured in both groups include perceived maternal self-efficacy, maternal infant bonding, and maternal depression after childbirth. A qualitative descriptive design will be used in phase two. Semi-structured interviews will be conducted with the participants to explore their experiences of the AT. Descriptive analysis, independent sample t-test, paired sample t-test, and regression analysis will be used for analysis of the quantitative data in phase one. Qualitative data from phase two will be analysed using thematic analysis.

Findings of this study may provide evidence on the use of AT to cope with FOC during pregnancy. If proven to be beneficial, AT may potentially be introduced and advocated as an intervention for women with FOC.

DETAILED DESCRIPTION:
Research Design:

A mixed-methods sequential explanatory design will be used. Phase one will be quasi-experimental study design, comparing women with FOC who received art therapy (experimental group) and women who received routine antenatal care (control group). A qualitative descriptive design will be used in phase two to explore the experiences of the participants who had art therapy for FOC.

Sampling:

Convenience sampling will be used for phase one. Purposive sampling will be used for phase two, for which only participants who had undergone the art therapy intervention will be invited to participate.

Consented participants will be invited to fill in the Fear of Birth Scale (FOBS). Participants with FOBS score of 60 and above will be enrolled into the study. Participants will be invited to participate in the Art Therapy intervention (experimental group). If participants are not agreeable to participate in the art therapy, they will be allocated to the control group.

Participants who had undergone the Art Therapy intervention will be invited to participate in phase two.

Sample Size:

Phase One: The study team is targeting to recruit 1200 participants to screen for FOC in phase one. Participants with FOC will be invited to continue participation in the quasi-experimental study with a target allocation of 1:1 in each group.

Phase Two: The sample size will be determined by data saturation, whereby no new information is identified from the data. This is estimated to be about sample size of 30 participants.

Data Collection Procedures:

Phase One:

Potential participants who are in the second trimester of their pregnancy (between 13 and 27 weeks of gestation) will be approached in the antenatal clinics. Details of the study will be explained using the Participant Information Sheet (PIS). After which, the FOBS will be used to measure the FOC. Recruited participants will be asked to fill in a hardcopy questionnaire.

After the participant has completed the questionnaire, the FOBS score will be tabulated and participants with FOBS score of more than or equal to 60 will be invited to participate in the intervention, which is a series of three to five art therapy sessions, depending on the participants' needs/preferences.

Women who are willing to participate in the art therapy sessions will be included in the experimental group, while women who received routine antenatal care but are not agreeable to participate in the art therapy sessions will be included in the control group. A study team member will contact the participants to arrange for the art therapy sessions and administration of the questionnaires.

A set of art materials will be provided to participants to use throughout the art therapy sessions, and to encourage participants to continue artmaking for self-care outside of sessions. The first session will be in a face-to-face format at a date and time agreed by the participant. Subsequent sessions will be offered via telehealth on dates and times agreed by the participant. Each session will last between 60 to 90 minutes and will be facilitated by an Art Therapist. Each session will be structured around themes aimed at building self-awareness, encouraging expressions of difficult emotions, strengthening the bond between participants and their child, and to facilitate the verbal counselling within the safety of art therapy session. FOBS score will be obtained from all the participants again in both experimental group and control group between 37 and 40 weeks of gestation in the form of hard copy questionnaire. Study procedures will be stopped for participants who delivered before the completion of the second administration of FOBS.

Participants in both experimental and control group will be contacted again at 1 month after childbirth. PMPS-E, PBQ, and EPDS will be administered. Participants will be provided with a link to access the online questionnaire.

Phase Two:

The first 30 participants who had undergone the art therapy sessions will be invited to participate in the individual semi-structured interviews. Interviews will be conducted face-to-face in a quiet and conducive room, or through phone call at 1 month after birth.

Interviews will be audio-recorded with permission from the participant and transcribed verbatim. The interview will be conducted by a trained midwife who is not involved in the art therapy sessions or the childbirth process of the participant.

Data Analysis:

Phase One: The following statistical analyses will be used. A value of p<0.05 will be assumed for the level of significance.

* Descriptive analysis will be used to describe the socio-demographic characteristics and all outcome variables (FOBS, PMPS-E, PBQ, and EPDS scores).
* Chi-squared test will be used to compare proportions of mode of birth and usage of epidural during labour between the experimental and control group.
* Paired sample t-test to compare the FOBS scores in the experimental group before and after intervention.
* Paired sample t-test to compare the FOBS scores in the control group in the second trimester and 37-40 weeks of pregnancy.
* Chi-squared test will be used to compare the number of pregnant women whose FOBS score decreased from ≥ 60 to a score less than 60 in both groups.
* Independent sample t-test will be used to compare all outcome variables (post FOBS, PMPS-E, PBQ, and EPDS scores) between the experimental and control groups.
* Pearson correlation analysis will be done to determine the associations between FOBS score and PMPS-E, PBQ, and EPDS scores of all participants.
* Pearson correlation analysis will be done to determine the associations between FOBS score and the socio-demographic variables.
* Univariate analysis will be done to compare the socio-demographic variables between the experimental and control groups.
* Regression analysis will be used to determine the predictors for FOC using the cut-off point for FOC (FOBS ≥ 60)

Phase Two:

Qualitative data will be analysed using thematic analysis, whereby data will be examined to identify common themes.

ELIGIBILITY:
Phase I

Inclusion Criteria:

1. Aged between 21 and 50 years old
2. English literate
3. Having an intrauterine singleton live pregnancy
4. Currently in the second trimester of the pregnancy (between 13 to 27 weeks of pregnancy)
5. Fear of Birth Scale (FOBS) score of 60 and above

Exclusion Criteria:

1. With contraindication for vaginal birth (for example placenta covering cervix)
2. With obstetric complications during pregnancy such as fetal anomaly that is incompatible with life
3. With current depression requiring medical intervention
4. Who had stillborn delivery

Phase II Inclusion Criteria Enrolled participants who had undergone the Art Therapy intervention in phase one

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females will be included in this study.
Enrollment: 100 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Fear or Childbirth (FOC) | From Screening (Second Trimester) to between 37 and 40 Weeks of Gestation
  FOC is measured by the Fear of Birth Scale (FOBS). The FOBS score ranges from 0 to 100. A higher score represents a higher value of fear of childbirth.

SECONDARY OUTCOMES:
Perceived Maternal Self-efficacy | Measured after study intervention period, one month after childbirth
  The Perceived Maternal Parental Self-Efficacy (PMPS-E) scale is a self-reported questionnaire to assess maternal parenting self-efficacy among postpartum women. It consists of 20 items theorized from four subscales.
  The PMPS-E scale ranges from 20 to 80. A higher score represents a higher level of maternal self-efficacy.
Maternal Infant Bonding | Measured after study intervention period, one month after childbirth
  The Postpartum Bonding Questionnaire (PBQ) is a self-reported questionnaire consisting of 25 items to measure maternal infant bonding with four factors, namely general emotional factor, anger towards and rejection of baby, infant-focus anxiety, and risk of abuse. Total score ranges from 0 to 125, with higher values indicating more bonding difficulties.
Maternal Depression after Childbirth | Measured after study intervention period, one month after childbirth
  The Edinburgh Postnatal Depression Scale (EPDS) is a self-reported questionnaire consisting of 10 items assessing symptoms of depression in the past week. There are four possible responses scored on a scale from 0 to 3. The total score is generated by summation of all items and ranges from 0 to 30.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Qi Ang, MSc(Nursing), Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams SS, Eberhard-Gran M, Eskild A. Fear of childbirth and duration of labour: a study of 2206 women with intended vaginal delivery. BJOG. 2012 Sep;119(10):1238-46. doi: 10.1111/j.1471-0528.2012.03433.x. Epub 2012 Jun 27. PMID 22734617
- [Background] Alehagen S, Wijma B, Wijma K. Fear of childbirth before, during, and after childbirth. Acta Obstet Gynecol Scand. 2006;85(1):56-62. doi: 10.1080/00016340500334844. PMID 16521681
- [Background] Alipour Z, Lamyian M, Hajizadeh E. Anxiety and fear of childbirth as predictors of postnatal depression in nulliparous women. Women Birth. 2012 Sep;25(3):e37-43. doi: 10.1016/j.wombi.2011.09.002. Epub 2011 Sep 29. PMID 21959041
- [Background] Barnes CR, Adamson-Macedo EN. Perceived Maternal Parenting Self-Efficacy (PMP S-E) tool: development and validation with mothers of hospitalized preterm neonates. J Adv Nurs. 2007 Dec;60(5):550-60. doi: 10.1111/j.1365-2648.2007.04445.x. PMID 17973719
- [Background] Brockington IF, Fraser C, Wilson D. The Postpartum Bonding Questionnaire: a validation. Arch Womens Ment Health. 2006 Sep;9(5):233-42. doi: 10.1007/s00737-006-0132-1. Epub 2006 May 4. PMID 16673041
- [Background] Challacombe FL, Nath S, Trevillion K, Pawlby S, Howard LM. Fear of childbirth during pregnancy: associations with observed mother-infant interactions and perceived bonding. Arch Womens Ment Health. 2021 Jun;24(3):483-492. doi: 10.1007/s00737-020-01098-w. Epub 2020 Dec 17. PMID 33336315
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Haines HM, Pallant JF, Fenwick J, Gamble J, Creedy DK, Toohill J, Hildingsson I. Identifying women who are afraid of giving birth: A comparison of the fear of birth scale with the WDEQ-A in a large Australian cohort. Sex Reprod Healthc. 2015 Dec;6(4):204-10. doi: 10.1016/j.srhc.2015.05.002. Epub 2015 May 15. PMID 26614602
- [Background] Hildingsson I, Rubertsson C. Depressive symptoms during pregnancy and after birth in women living in Sweden who received treatments for fear of birth. Arch Womens Ment Health. 2022 Apr;25(2):473-484. doi: 10.1007/s00737-022-01213-z. Epub 2022 Feb 21. PMID 35190877
- [Background] Hildingsson I, Rubertsson C. Postpartum bonding and association with depressive symptoms and prenatal attachment in women with fear of birth. BMC Pregnancy Childbirth. 2022 Jan 25;22(1):66. doi: 10.1186/s12884-021-04367-3. PMID 35078403
- [Background] Kinsella MT, Monk C. Impact of maternal stress, depression and anxiety on fetal neurobehavioral development. Clin Obstet Gynecol. 2009 Sep;52(3):425-40. doi: 10.1097/GRF.0b013e3181b52df1. PMID 19661759
- [Background] Nieminen K, Stephansson O, Ryding EL. Women's fear of childbirth and preference for cesarean section--a cross-sectional study at various stages of pregnancy in Sweden. Acta Obstet Gynecol Scand. 2009;88(7):807-13. doi: 10.1080/00016340902998436. PMID 19488882
- [Background] Nilsson C, Hessman E, Sjoblom H, Dencker A, Jangsten E, Mollberg M, Patel H, Sparud-Lundin C, Wigert H, Begley C. Definitions, measurements and prevalence of fear of childbirth: a systematic review. BMC Pregnancy Childbirth. 2018 Jan 12;18(1):28. doi: 10.1186/s12884-018-1659-7. PMID 29329526
- [Background] O'Connell MA, Leahy-Warren P, Khashan AS, Kenny LC, O'Neill SM. Worldwide prevalence of tocophobia in pregnant women: systematic review and meta-analysis. Acta Obstet Gynecol Scand. 2017 Aug;96(8):907-920. doi: 10.1111/aogs.13138. Epub 2017 May 17. PMID 28369672
- [Background] O'Connor TG, Heron J, Golding J, Beveridge M, Glover V. Maternal antenatal anxiety and children's behavioural/emotional problems at 4 years. Report from the Avon Longitudinal Study of Parents and Children. Br J Psychiatry. 2002 Jun;180:502-8. doi: 10.1192/bjp.180.6.502. PMID 12042228
- [Background] Raisanen S, Lehto SM, Nielsen HS, Gissler M, Kramer MR, Heinonen S. Fear of childbirth predicts postpartum depression: a population-based analysis of 511 422 singleton births in Finland. BMJ Open. 2013 Nov 28;3(11):e004047. doi: 10.1136/bmjopen-2013-004047. PMID 24293208
- [Background] Rondung E, Thomten J, Sundin O. Psychological perspectives on fear of childbirth. J Anxiety Disord. 2016 Dec;44:80-91. doi: 10.1016/j.janxdis.2016.10.007. Epub 2016 Oct 18. PMID 27788373
- [Background] Slade P, Balling K, Sheen K, Houghton G. Establishing a valid construct of fear of childbirth: findings from in-depth interviews with women and midwives. BMC Pregnancy Childbirth. 2019 Mar 18;19(1):96. doi: 10.1186/s12884-019-2241-7. PMID 30885153
- [Background] Talge NM, Neal C, Glover V; Early Stress, Translational Research and Prevention Science Network: Fetal and Neonatal Experience on Child and Adolescent Mental Health. Antenatal maternal stress and long-term effects on child neurodevelopment: how and why? J Child Psychol Psychiatry. 2007 Mar-Apr;48(3-4):245-61. doi: 10.1111/j.1469-7610.2006.01714.x. PMID 17355398